CLINICAL TRIAL: NCT01385696
Title: Study Evaluating Preference, Satisfaction and Ease of Use of Inhalers in COPD Diagnosed Patients
Brief Title: Study Evaluating Preference, Satisfaction and Ease of Use of Inhalers in Chronic Obstructive Pulmonary Disease (COPD) Diagnosed Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Almirall, S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: M/34273/32
Record Dates: First submitted 2011-06-17; First posted 2011-06-30 (Estimated); Results first posted 2013-04-22 (Estimated); Last update posted 2015-06-24 (Estimated); Status verified 2015-05

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

ARMS (2):
- group A (Experimental): Genuair first, HandiHaler second
  Interventions: Device: Genuair® (Almirall S.A.); Device: HandiHaler® (Boehringer Ingelheim's)
- group B (Experimental): HandiHaler first, Genuair second
  Interventions: Device: Genuair® (Almirall S.A.); Device: HandiHaler® (Boehringer Ingelheim's)

INTERVENTIONS:
Device: Genuair® (Almirall S.A.) — Inhaler with only placebo, once daily, 14 days
Device: HandiHaler® (Boehringer Ingelheim's) — Inhaler with only placebo, once daily, 14 days

SUMMARY:
Preference study: Genuair vs HandiHaler inhalers in COPD patients.

ELIGIBILITY:
Inclusion Criteria:

* Adult male or female patients aged ≥ 40 with stable COPD
* Naïve patients to the use of study inhalers
* Patients agreeing on participating and signing the Informed Consent Form

Exclusion Criteria:

* Patients with other clinically significant disease, particularly body malformations or diseases affecting coordination and/or motor system
* Patients unable to read product package instructions and answer patient reported questionnaires

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2011-06; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jordi Estruch, Head of GMA, Study Director — Almirall, S.A.
Locations (4):
- Germany (2):
  - Almirall investigative site 3, Bonn
  - Almirall investigative site 5, Koblenz
- Netherlands (2):
  - Almirall investigative site 1, Enschede
  - Almirall investigative site 2, Zutphen

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted 4 centres, 2 in The Netherlands and 2 in Germany. The first patient was screened in June 2011 and the last patient visit was in January 2012.
Groups:
- Placebo Genuair (Daily) Then Placebo HandiHaler (Daily): Each morning, patients used the Genuair® (Almirall S.A.) inhaler containing placebo followed by the HandiHaler® (Boehringer Ingelheim) inhaler containing placebo. The study period consisted of 1 period of 14 days.
- Placebo HandiHaler (Daily) Then Placebo Genuair (Daily): Each morning, patients used the HandiHaler® (Boehringer Ingelheim) inhaler containing placebo followed by the Genuair® (Almirall S.A.) inhaler containing placebo. The study period consisted of 1 period of 14 days.
Period: Overall Study
Arm/Group | Placebo Genuair (Daily) Then Placebo HandiHaler (Daily) | Placebo HandiHaler (Daily) Then Placebo Genuair (Daily)
Started | 66 | 64 (1 patient used Handihaler® once only, Genuair® zero times, & was excluded from the safety population)
Completed | 66 | 64
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Overall Study Safety Population: All patients randomized into the study excluding 1 patient who used Handihaler® once only, Genuair® zero times, & was excluded from the safety population
Arm/Group | Overall Study Safety Population
Number analyzed (Participants) | 129
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.9 (8.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42
  Male | 87
Region of Enrollment [Number; unit: participants]
  Germany | 85
  Netherlands | 44

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients Who Prefer Genuair Device Versus Handihaler Device at Visit 2
Description: Patients will be asked to answer which device they prefer after 2 weeks of daily practice (visit 2)
Time Frame: 14 days
Population: ITT: all randomized patients who used both devices at least once and expressed a preference for either or neither inhaler. 24 patients (12 each arm) received the incorrect treatment allocation and were excluded from the ITT population. Missing data was handled via the observed cases approach.
Measure: Number; unit: Percentage of Patients
Groups:
- Overall Intention-to-treat Population: Overall intention-to-treat (ITT) population
Arm/Group | Overall Intention-to-treat Population
Number analyzed (Participants) | 105
Percentage of Patients
  Prefer Genuair inhaler | 68.6
  Prefer Handihaler inhaler | 18.1
  No preference | 13.3

2. Secondary Outcome: Mean Overall Satisfaction With Genuair and Handihaler at Visit 2
Description: The patient will be asked to rate the overall satisfaction with each device using a Likert-type scale (from 1 [very dissatisfied] to 5 [very satisfied]) after 2 weeks of daily practice (visit 2)
Time Frame: 14 days
Population: ITT: all randomized patients who used both devices at least once and expressed a preference for either or neither inhaler. 24 patients from the safety population (12 each arm) received the incorrect treatment allocation and were excluded from the ITT population. Missing data were handled via the observed cases approach.
Measure: Mean (95% Confidence Interval); unit: Units on a scale (1-5)
Groups:
- Genuair Inhaler; Handihaler Inhaler: Intention-to-treat (ITT) population
Arm/Group | Genuair Inhaler | Handihaler Inhaler
Number analyzed (Participants) | 104 | 105
Units on a scale (1-5) | 4.5655 [4.3132 to 4.8177] | 3.7944 [3.5425 to 4.0462]

3. Secondary Outcome: Percentage of Patients Making at Least 1 Critical Error Using the Genuair and Handihaler Devices at Visit 2
Description: The correct use of devices will be assessed measuring the errors made by patients when using each device after 2 weeks of daily practice (visit 2).
  Critical error is defined as the one that compromise the potential benefit of the treatment such as those that impede drug deposition in the lungs or delivery of sufficient dose.
Time Frame: 14 days
Population: as for outcome 2
Measure: Number; unit: Percentage of Patients
Arm/Group | Genuair Inhaler | Handihaler Inhaler
Number analyzed (Participants) | 104 | 105
Percentage of Patients | 10.5 | 26.7

ADVERSE EVENTS:
Groups:
- Genuair Then HandiHaler: The study period consisted of 1 period of 14 days. Every morning patients used the Genuair® (Almirall S.A.) inhaler containing placebo follow by the HandiHaler® (Boehringer Ingelheim) inhaler containing placebo.
- HandiHaler Then Genuair: The study period consisted of 1 period of 14 days. Every morning patients used the HandiHaler® (Boehringer Ingelheim)inhaler containing placebo follow by the Genuair® (Almirall S.A.) inhaler containing placebo.
Arm/Group | Genuair Then HandiHaler | HandiHaler Then Genuair
Serious Adverse Events (participants affected / at risk) | 0/66 | 0/63
Other Adverse Events (participants affected / at risk) | 0/66 | 0/63

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All the information related to this clinical trial is considered strictly confidential and is the property of Almirall. This information will not be given to a third party without the written consent of Almirall. Publication and/or presentation, whether complete or partial, of any part of the data or results of this trial will be subject to revision and written agreement between the investigator and Almirall.